CLINICAL TRIAL: NCT02052791
Title: An Open-label Study to Assess the Safety and Tolerability of ISIS 396443 in Patients With Spinal Muscular Atrophy Who Previously Participated in 396443-CS2 or 396443-CS10
Brief Title: An Open-label Safety and Tolerability Study of Nusinersen (ISIS 396443) in Participants With Spinal Muscular Atrophy (SMA) Who Previously Participated in ISIS 396443-CS2 (NCT01703988) or ISIS 396443-CS10 (NCT01780246)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 396443-CS12
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS 396443; IONIS-SMNRx; IONIS-SMN Rx; Spinraza
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nusinersen (Experimental)
  Interventions: Drug: nusinersen

INTERVENTIONS:
Drug: nusinersen — Administered by intrathecal (IT) injection
  Other Names: ISIS 396443; Spinraza; BIIB058; IONIS SMN Rx; ISIS SMNRx

SUMMARY:
The primary objective of this study is to examine the safety and tolerability of nusinersen (ISIS 396443) administered intrathecally to participants with Spinal Muscular Atrophy (SMA) who previously participated in ISIS 396443-CS2 (NCT01703988) or ISIS 396443-CS10 (NCT01780246). The secondary objective is to examine the plasma and cerebrospinal fluid (CSF) pharmacokinetic(s) (PK) of nusinersen administered intrathecally to participants with SMA who previously participated in ISIS 396443-CS2 or ISIS 396443-CS10.

DETAILED DESCRIPTION:
This study was conducted and the protocol was registered by Ionis Pharmaceuticals, Inc.

In August 2016, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical signs attributable to Spinal Muscular Atrophy
* Satisfactory completion of dosing and all study visits in ISIS 396443-CS2 (NCT01703988) or ISIS 396443 CS10 (NCT01780246) with an acceptable safety profile, per Investigator judgement.
* Able to complete all study procedures, measurements and visits and parent/participant has adequately supportive psychosocial circumstances, in the opinion of the investigator
* Estimated life expectancy > 2 years from Screening
* Meets age-appropriate institutional criteria for use of anesthesia/sedation, if use is planned for study procedure

Key Exclusion Criteria:

* Have any new or worsening of existing condition which in the opinion of the Investigator would make the subject unsuitable for enrollment, or could interfere with the participant participating in or completing the study.
* Dosing in ISIS 396443-CS2 (NCT01703988) or ISIS 396443-CS10 (NCT01780246) within 180 days (6 months) of screening, or longer ago than 396 days (13 months) from screening
* Hospitalization for surgery (i.e. scoliosis surgery) or pulmonary event within 2 months of screening or planned during the duration of the study
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy
* Clinically significant abnormalities in hematology or clinical chemistry parameters
* Treatment with another investigational drug, biological agent, or device within 1-month of Screening or 5 half-lives of study agent, whichever is longer. Any history of gene therapy or cell transplantation.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events | Up to 24 Months
Number of participants with clinically significant neurological examination abnormalities | Up to 24 Months
Number of participants with clinically significant vital sign abnormalities | Up to 24 Months
Number of participants with clinically significant physical examination abnormalities | Up to 24 Months
Number of participants with clinically significant weight abnormalities | Up to 24 Months
Number of participants with clinically significant laboratory parameters | Up to 24 Months
Number or participants with clinically significant cerbrospinal fluid (CSF) laboratory parameters | Up to Day 176
Number of participants with clinically significant electrocardiograms (ECGs) abnormalities | Up to 24 Months
Change from Baseline in concomitant medications | Up to 24 Months

SECONDARY OUTCOMES:
PK parameters of nusinersen (ISIS 396443) in CSF levels: Maximum observed plasma drug concentration (Cmax) | Pre-dose Day 176, Day 358 and Day 540
PK parameters of nusinersen in CSF levels: Time to reach maximum observed concentration (Tmax) | Pre-Dose Day 176, Day 358 and Day 540
PK parameters of nusinersen in CSF levels: Area under the plasma concentrations time curve from the time of the intrathecal (IT) dose to the last collected sample (AUCinf) | Pre-Dose Day 176, Day 358 and Day 540

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - UT Southwestern Medical Center - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Derived] Darras BT, Farrar MA, Mercuri E, Finkel RS, Foster R, Hughes SG, Bhan I, Farwell W, Gheuens S. An Integrated Safety Analysis of Infants and Children with Symptomatic Spinal Muscular Atrophy (SMA) Treated with Nusinersen in Seven Clinical Trials. CNS Drugs. 2019 Sep;33(9):919-932. doi: 10.1007/s40263-019-00656-w. PMID 31420846
- [Derived] Darras BT, Chiriboga CA, Iannaccone ST, Swoboda KJ, Montes J, Mignon L, Xia S, Bennett CF, Bishop KM, Shefner JM, Green AM, Sun P, Bhan I, Gheuens S, Schneider E, Farwell W, De Vivo DC; ISIS-396443-CS2/ISIS-396443-CS12 Study Groups. Nusinersen in later-onset spinal muscular atrophy: Long-term results from the phase 1/2 studies. Neurology. 2019 May 21;92(21):e2492-e2506. doi: 10.1212/WNL.0000000000007527. Epub 2019 Apr 24. PMID 31019106
- See also: Cure SMA — http://www.curesma.org
- See also: Muscular Dystrophy Association — http://mda.org/disease/spinal-muscular-atrophy
- See also: National Organization for Rare Diseases — https://www.rarediseases.org
- See also: Clinical Study Report (CSR) Synopsis - a results summary — http://clinicalresearch.biogen.com/Content/Studies/CS12%20Biogen.com%20Packet.pdf